CLINICAL TRIAL: NCT05114135
Title: First-in-man Safety and Performance of OSTEO3 ZP PUTTY in Subjects Undergoing Transforaminal Lumbar Interbody Fusion
Brief Title: TLIF Osteo3 ZP Putty Study (Also Known as the TOP Fusion Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OssDsign (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIR202001
Record Dates: First submitted 2021-09-09; First posted 2021-11-09 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Lumbar Spinal Stenosis
Keywords: synthetic bone graft, TLIF, Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: 40-65-year-old adults requiring one level instrumented spine fusion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject group (Experimental): undergoing instrumented TLIF with instrumented PLF using investigational product as synthetic bone graft
  Interventions: Device: Osteo3 ZP Putty

INTERVENTIONS:
Device: Osteo3 ZP Putty — Transforminal Interbody Fusion at one spinal level (L2-S1) with instrumented posteriorlateral fusion on at least the contralateral side to the TLIF approach.
  Other Names: OssDsign Catalyst

SUMMARY:
In recent years there has been an increase in interest from surgeons in the use of synthetic bone graft substitutes to avoid the need of sourcing allograft or iliac crest autograft for use in spinal fusion procedures. This will be an open label, prospective, first in man, single-centre clinical study to evaluate the safety and performance of Osteo3 ZP Putty synthetic bone graft in TLIF procedures with instrumented PLF. Safety and performance data obtained in this clinical study will be used to estimate clinical success rates achieved with the use of Osteo3 ZP Putty synthetic bone graft in TLIF procedures. No comparative control group is intended.

The study is expected to run for approximately three years with each subject being followed up for a two- year post-operative period. The target is to recruit approximately 17 subjects to this clinical study, allowing for some subject attrition to get 15 evaluable.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with DDD (as defined below), degenerative spondylolisthesis or lumbar spinal stenosis at one spinal level:

DDD defined as one or more of the following: instability as defined by greater than or equal to 3 mm translation or greater than or equal to 5 degrees angulation, decreased disc height, on average by greater than or equal to 2 mm, but dependent upon the spinal level, scarring/thickening of ligamentum flavum or annulus fibrosis, herniated nucleus pulposus or vacuum phenomenon.

* The subject has failed at least six months of non-operative treatment prior to clinical study enrolment (e.g. bed rest, physical therapy, bracing, traction, drug therapy, etc) and is a candidate for spinal fusion surgery over one vertebral level between, and including, L2 to S1 (i.e. second lumbar to first sacral).
* The subject is 40-65 years old.
* The subject is, in the Investigator's opinion, psychosocially healthy and physically able to fully comply with this protocol, including the post-operative regimen, required follow up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

* Subject has diagnosis of symptomatic DDD, spondylolisthesis, or lumbar spinal stenosis at more than one level.
* Subject has had prior surgery at any lumbar level.
* Subject has systemic infection or infection at the surgical site.
* History of significant metabolic bone disease such as osteomalacia, autoimmune disease including rheumatoid arthritis, renal disease, hepatic disease, peripheral vascular disease, insulin dependent diabetes, Paget's disease at the involved spinal level(s) or upper motor neuron disease (positive Babinski sign).
* Subject has a medical condition that would interfere with post-operative assessments and care (i.e. psychiatric disease, paraplegia, quadriplegia, etc.).
* Subject is in poor general health or any concurrent disease process that would place the subject in excessive risk to surgery (e.g. significant circulatory, pulmonary problems, or cardiac disease).
* Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the Investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow up.
* The subject is known to be pregnant/breastfeeding at the time of enrolment or plans to become pregnant during their participation in the clinical study.
* Subject is participating in, or has completed within the last 30 days, another investigational clinical study, which could confound results.
* Morbid obesity defined as a Body Mass Index (BMI) ≥ 40.
* Has or has had a tumour or fracture at the involved level.
* Subject has a condition or requires post-operative medications that may interfere with bone/soft tissue healing (i.e. NSAIDS, oral or parenteral glucocorticoids, immunosuppressants, methotrexate, etc.), or that effect the rate of bone metabolism unless they have undergone a 14 day wash out period prior to surgery.
* Subject is taking medication for treatment of osteoporosis and/or in the Investigator's opinion, spinal instrumentation would be contraindicated.
* Subject has a T-score of less than -2.5 is therefore diagnostic of osteoporosis.
* Subject is involved in on-going litigation concerning their medical condition.
* Subject has a known allergy to silicon.
* Long-term use (longer than 3 months) of opiates.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of device-related serious adverse events | 24 months
  Incidence of device-related serious adverse events. Success measured as no treatment-related events occurring in 24 months post-surgery.
Percentage of subjects with evidence of interbody fusion being achieved in 12 months post-surgery | 12 months
  Percentage of subjects with evidence of interbody fusion being achieved in 12 months post-surgery. Assessed as any evidence of bridging bone observed joining the superior and inferior vertebral bodies. Scored using a simple scoring of yes, no or not known if cannot be seen.

SECONDARY OUTCOMES:
Oswestry Disability Index questionnaire to assess Quality of life | 3,6,12 and 24 months (unless fused at 12 months)
  Validated off-the-shelf questionnaire asking patients questions about their ability to perform basic life tasks. It will be used to assess both the subject's back pain and how that pain affects the subject's ability to manage in everyday life. The questionnaire is divided into ten sections designed to assess limitations of various activities of daily living. Each section contains six statements and each statement describes a greater degree of difficulty in that activity than the preceding statement. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The scores for all sections are added together, giving a possible score of 50. The total is doubled and expressed as a percentage.
Visual Analog Score to measure pain | 3,6,12 and 24 months (unless fused at 12 months)
  Subject will score their pain from 0 to 100 by making a mark on a 10cm line where 0 = no pain and 100 = worst pain imaginable. The change in score from baseline (pre-surgical score) will be assessed at the time points below and reported as a percentage change.
SF-36 short form to assess change in how the subjects back pain has affected their quality of life. | 3,6,12 and 24 months (unless fused at 12 months)
  It will be used to assess both the subject's back pain and how that pain affects the subject's ability to manage in everyday life. The questionnaire is divided into eleven sections designed to assess limitations of various activities of daily living. Subject will score each section and the resulting scores are entered into a validated software evaluation tool which produces a result out of 100, allowing percentage change to be assessed from baseline (pre-surgical) score. Change in score will be assessed at the time points below and reported as a percentage change.
Maintenance or Improvement in Neurological function | 3,6,12 and 24 months (unless fused at 12 months)
  The subject will be assessed for neurological function by physical examination. Success = maintenance or improvement in neurological function compared to baseline scores for all Neurological assessments described as separate outcome measures below (Outcome measures 9 - 14 below). Subject will be considered to have clinical success if all neurological outcomes (outcomes 9-14) are maintained or improved from baseline assessments.
Safety: Incidence rate and type of device-related Adverse events | 24 months
  Incidence rate and type of device-related Adverse events (AEs) recorded will be described for the 24 months post surgery period
Bone Fusion Success | 3, 6 and 24 months
  Presence of bone fusion assessed by CT scans at 3, 6 months and 24 months. Scored as yes or no for presence of a bridge of bone between the superior and inferior vertebral bodies. The results will be reported as percentage of subjects fused at the various timepoints below.
Neurological outcome - Maintenance or improvement of sensory response at dermatomal levels operated in each leg when compared to baseline scores | 3,6,12 and 24 months (unless fused at 12 months)
  Sensory - Decreased sensation will be assessed by evaluating sensation response (e.g., to pin prick, light touch or vibration) for the involved dermatomal levels. The examination method chosen to make these assessments will be left to the discretion of the Investigator. Sensory function will be scored as 0 = Absent, 1 = Impaired, 2 = Normal
Neurological outcome - Maintenance or improvement in patellar and Achilles deep tendon reflexes in each leg when compared to baseline scores | 3,6,12 and 24 months (unless fused at 12 months)
  Reflex - Reflexes of both legs will be evaluated by assessing patellar (knee jerk) and Achilles (ankle jerk) deep tendon reflexes. The Investigator will be asked to indicate whether the knee and ankle reflex response for each leg is normal, decreased, absent or increased.
Neurological outcome - Maintenance or improvement of muscle strength at all muscle sites assessed in each leg when compared to baseline scores | 3,6,12 and 24 months (unless fused at 12 months)
  Muscle Strength - Muscle strength of both legs will be assessed bilaterally at the following muscle sites: hip flexors (iliopsoas musculature); knee extensors (quadriceps); ankle dorsiflexors (tibialis transforaminal); ankle plantar flexors (gastrocnemius); and long toe extensors (extensor halluces longus) using the following clinical scale. The worst assessment (no evidence of contractility) will be assigned the lowest clinical score 0 out of 5 while full range of motion against gravity, full resistance will be assigned the highest clinical score 5 out of 5. The following scale will be used to assess muscle strength:
  No evidence of contractility 0 Slight contractility, no movement 1 Full range of motion, gravity eliminated (passive movement) 2 Full range of motion with gravity 3 Full range of motion against gravity, some resistance 4 Full range of motion against gravity, full resistance 5
Neurological outcome - Maintenance of a negative straight leg raising response or improvement of a positive straight leg raising response to negative in each leg when compared to the baseline result. | 3,6,12 and 24 months (unless fused at 12 months)
  Straight Leg Raising - The ability of the subject to undergo passive straight leg raising manoeuvres while in the supine position will be assessed for both legs. The results will be recorded as a positive or negative straight leg raise (SLR) for each leg.
Neurological outcome - Maintenance of a negative femoral stretch response or improvement of a positive femoral stretch response to negative in each leg when compared to the baseline result | 3,6,12 and 24 months (unless fused at 12 months)
  Femoral Stretch - The ability of the subject to undergo passive femoral stretch manoeuvres while lying on one side will be assessed for both legs. The results will be recorded as a positive or negative femoral stretch for each leg.
Absence of Babinski's sign | 3,6,12 and 24 months (unless fused at 12 months)
  Presence or absence of Babinski's sign will be recorded. Absence of Babsinki's sign is considered normal and a success.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Varga, MD, Principal Investigator — National Spine Centrer, Buda Health Center, Budapest
Locations (1):
- Buda Health Center, Királyhágó u. 1-3., Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available